CLINICAL TRIAL: NCT05896124
Title: A Phase II Study to Evaluate Safety, Tolerability and Efficacy, of CS0159 in Patients Subjects With PBC (Primary Biliary Cholangitis), Multicenter, Randomized 12-week, Double-blind, Placebo-controlled, and 40-weeks Open Study
Brief Title: CS0159 in Chinese Patients With PBC (Primary Biliary Cholangitis)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBC-CS0159-004
Record Dates: First submitted 2023-05-17; First posted 2023-06-09 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2mg CS0159 (Experimental): QD for 12 weeks
  Interventions: Drug: 2mg CS0159; Drug: Placebo
- 4mg CS0159 (Experimental): QD for 12 weeks
  Interventions: Drug: 2mg CS0159
- Placebo (Experimental): QD for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2mg CS0159 — Oral QD
  Arms: 2mg CS0159; 4mg CS0159
Drug: Placebo — Oral QD
  Arms: 2mg CS0159; Placebo

SUMMARY:
A phase II study to evaluate safety, tolerability and efficacy of CS0159 in patients with PBC (Primary Biliary Cholangitis).

DETAILED DESCRIPTION:
This is a phase II study to evaluate safety, tolerability and efficacy of CS0159 in patients with PBC (Primary Biliary Cholangitis). The study has been designed to have two parts, the first part of the study will be double-blinded for 12 weeks. The second part of the study will be an open-label trail lasting 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. When signing ICF age≥18 years≤75 years, male or female
2. Meets the diagnostic criteria of PBC, such as elevation ALP, positive AMA or AMA-M2, If negative for AMA, positive for PBC specific antibody and Liver biopsy meeting PBC criteria six months before screening
3. 1.67 × ULN ≤ALP ≤ 10 × ULN and TBil≤ 3 × ULN
4. UDCA≥6 months before randomization and a stable dose (no less than 13-15 mg/kg/d in principle) ≥3 months after the efficacy was poor (meeting inclusion criteria 3), or UDCA was not tolerated, and stop taking UDCA (no UDCA use for ≥3 months before randomization)
5. Understand the study content, comply with the study protocol, and sign the ICF voluntarily

   -

Exclusion Criteria:

1. ALT or AST>5×ULN；
2. OCA(Obercholic acid) in the 3 months prior to randomization
3. Known concomitant hepatobiliary disease or history
4. Significant hepatic impairment as defined by Child-Pugh classification of B or C, history of liver transplantation, current placement on a liver transplant list or current Model for End Stage Liver Disease (MELD) score ≥15.
5. Patients were screened for HBsAg positive, HCVAb positive, HIV Ab positive, or TPAb positive.
6. (creatinine, Cr) ≥1.5×ULN and Cr clearance rate <60 mL/min
7. Platelet<80×10^9/L；
8. INR>1.3
9. ALB<3.5 g/dL
10. Severe pruritus or systemic medication was required within 2 months prior to randomization
11. Arrhythmia, Or during screening the QTc interval was ≥450 ms for male and 470 ms for female
12. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolism in the large intestine, eg, inflammatory bowel disease, prior or planned (during the study period) bariatric surgery (such as gastroplasty, roux-en-Y gastric bypass).
13. Concomitant use of medications, food, and drinks that are strong or moderate CYP3A4 inhibitors or inducers within 14 days prior to the first dose of study drug and throughout the study duration.
14. Diseases that may cause non-hepatic elevation of ALP (such as Paget's disease) or may result in a life expectancy of less than 2 years
15. A history of malignant tumor within 5 years prior to randomization
16. Perazathioprine, colchicine, cyclosporine, methotrexate, mycophenolate, and pentoxifylline were administered from 28 days before randomization to the entire clinical study period. Fenofibrate or other Bates; Budesonide and other systemic corticosteroid hormones; Hepatotoxic drugs; Liver protection Drugs and other hepatoprotective drugs were given a stable dose <28 days before randomization or could not be maintained during the trial; cholagogue
17. The administration of interleukin or other cytokine antibodies, as well as chemical factors or immunotherapy, was prohibited from 12 months prior to randomization throughout the clinical study period
18. Substance abuse or alcoholism from 6 months prior to randomization throughout the entire clinical study period
19. Poor blood pressure control is indicated by a systolic pressure greater than 160 mmHg or diastolic pressure greater than 100 mmHg during screening
20. Poor blood glucose control, that is, HBA1c >9.0% at screening
21. Pregnancy, planned pregnancy, lactation
22. Use of other investigational drugs within 3 months
23. Any other condition(s) that would compromise the safety of the patient or compromise the quality of the clinical study, as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
AE incidence | baseline to 12 weeks
  AE incidence in three arms
relative changes from baseline in ALP at week 12 | baseline to 12 weeks
  Compared with placebo ,Percentage change of CS0159 to ALP relative to baseline

SECONDARY OUTCOMES:
Absulute changes from baseline in ALP at week 12 | baseline to 12 weeks
  Compared with placebo, CS0159 changes in serum ALP relative to baseline
ALP and TBil | baseline to 12 weeks
  Compared with placebo, the rate of subjects to achive the lelve of ALP< 1.67 ULN and (total bilirubin) TBil ≤ULN
Pruritus | from basline to 40 weeks
  the changes from baseline in Pruritus to week 40
Liver function: ALT, AST, ALB, LDL-C, HDL-C, TBA, GGT, TC, TG | from baseline to week 40.
  The reduction of ALT, AST, ALB, LDL-C, HDL-C, TBA, GGT, TC, and TG from baseline to week 40.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Deng, Study Director — Cascade Pharmaceuticals, Inc
Locations (16):
- China (16):
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Friendship Hospital, Captail Medcial University, Beijing, Beijing Municipality
  - Beijing Youan Hostital, Captial Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangzhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - The Seconed Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Shaoyifu Hospital of Zhejiang University Medical, Hangzhou, Zhejiang
  - The First Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang